CLINICAL TRIAL: NCT03979937
Title: Development and Validation of a Simple Diagnostic Tool Predictive of the Aseptic Character of Joint Effusion
Acronym: PRASEPT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier le Mans (Other)
Responsible Party: Sponsor
Other Study IDs: CHM-2019/S7/03
Record Dates: First submitted 2019-06-06; First posted 2019-06-10 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Joint Effusion; Septic Arthritis; Arthritis
MeSH Terms: conditions — Hydrarthrosis; Arthritis, Infectious; Arthritis | interventions — Arthrocentesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Arthrocentesis — Arthrocentesis to determine the nature of the effusion (septic or aseptic).

SUMMARY:
Development and validation of a simple diagnostic tool predictive of the aseptic character of joint effusion in the primary care setting.

DETAILED DESCRIPTION:
In accordance with guidelines and because of the potential gravity that this situation could represent, any joint effusion must be considered as a septic arthritis until proven otherwise, thus justifying an arthrocentesis and an adequate treatment. Nevertheless, because of epidemiology in primary care, this pragmatic attitude is quite commonly obscured and practices vary according to the experience of the doctor and his personal habits. As a result, the arthrocentesis is not commonly performed and anti-inflammatory treatment, whether based on NSAIDs or corticosteroids, is even sometimes administered to the patient despite the contrary guidelines. Although usually effective, this attitude is however not without risks. In this context, it seems interesting to develop a simple, reproducible and applicable diagnostic tool in a primary care setting for predicting the risk of septic arthritis.

This study is therefore aimed at the development and validation of a predictive score based on simple clinical and paraclinical data (such as the macroscopic appearance of the synovial fluid removed) in a patient with an effusion, whatever either the clinical presentation, whether isolated or integrated in a more complex clinical presentation, whether associated with locoregional inflammatory or general signs or not.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (age ≥ 18 years)
* Hospitalized in the conventional hospitalization unit or day hospitalization unit or received in consultation within the Rheumatology or Infectious Diseases units at the Le Mans General Hospital
* presenting at least one joint effusion at clinical examination
* Interesting a native, nonoperated joint, accessible to a puncture based on clinical markers, determined by palpatory anatomy
* Affiliated to social security
* No opposition expressed after written information

Exclusion Criteria:

* General antibiotic therapy in progress or completed less than 15 days before
* Failure to perform the arthrocentesis
* Person subject to a legal protection measure, not allowing his compliance with the study
* Participant already included in another study (exclusivity clause)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult patients presenting with at least one clinical joint effusion accessible to arthrocentesis, interesting a native non operated joint, without any general antibiotic therapy in the previous 15 days.
Sampling Method: Non-Probability Sample
Enrollment: 328 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Presence of a septic arthritis | 10 days after the arthrocentesis.
  Presence of more than 2000 cells/mL and bacterial growth in the articular fluid.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle Dernis, MD, Principal Investigator — Centre Hospitalier du Mans, Rheumatology Department
Locations (1):
- Centre Hospitalier Le Mans, Le Mans, France

IPD SHARING:
Plan to Share IPD: No